CLINICAL TRIAL: NCT04810871
Title: Surgical Resection of Latent Brain Tumors Prior to Recurrence
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: internal procedural reasons
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-013059; NCI-2021-01950 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-013059 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2021-03-15; First posted 2021-03-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (surgery) (Experimental): Patients undergo surgery as indicated clinically when applicable.
  Interventions: Procedure: Brain Surgery

INTERVENTIONS:
Procedure: Brain Surgery — Undergo surgery

SUMMARY:
This clinical trial evaluates the side effects and possible benefits of operating on brain tumors prior to the tumor coming back (recurrence). Understanding when surgery is most useful to patients with brain tumors is important. Some patients may undergo chemotherapy or radiation but still have visible tumor remaining after treatment. The purpose of this research is to compare outcomes of those who have surgery after chemotherapy or radiation, but prior to tumor recurrence, to those who have surgery at a different time, or no surgery at all.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and feasibility of surgical resection for pre-recurrent brain tumors.

SECONDARY OBJECTIVES:

I. To determine whether there are differences in overall survival for patients who receive radiation therapy (RT) prior to surgery as compared to patients who receive RT after surgery or patients undergoing no further surgery.

II. To determine for patients having pre-recurrent surgery whether there is a longer interval to local/regional progression, any central nervous system (CNS) progression or need for subsequent intracranial treatment compared to patients receiving post-operative RT, time to each will be separately documented.

III. To determine for patients with pre-operative as compared to post-operative fractionated radiation for brain metastases (mets) whether there is a decreased rate of local recurrence.

IV. To determine for patients with pre-operative as compared to post-operative fractionated radiation for brain mets whether there is a decreased rate of leptomeningeal disease.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine the genetic and molecular alterations occurring in radiated brain and radiated tumor tissue compared to nonradiated tissue specimens (subjects will be matched to Mayo Clinic Cancer Center Neuro-Oncology Program Registry for the study of Nervous System Tumors 12-003458).

II. To investigate the relative sensitivity of radiated human CNS tumors to senolytic or other therapies in ex vivo assays targeting radiation-induced biology to promote synthetic lethality using cryopreserved or fresh tissue.

III. To investigate the availability and utility of candidate biomarkers reflective of tumor burden and therapeutic susceptibility, from tissue, cerebrospinal fluid (CSF) and peripheral blood.

IV. Patients self-reported outcomes may be obtained through the Neurosurgery Registry program. As available, these data may be referenced as a screening tool for any impact on quality of life (QOL) associated with trial participation as compared to matched controls.

OUTLINE:

Patients undergo surgery as indicated clinically when applicable. Patients also undergo magnetic resonance imaging (MRI) or computed tomography (CT) throughout the study and may optionally undergo tissue sample collection on study.

After completion of surgery, patients are followed up at 3 and 6 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological or cytological confirmation of brain tumor and/or suspected brain tumor based on clinical and radiologic findings
* Prior chemotherapy and/or radiation treatment directed to the known/suspected tumor
* Radiographic evidence of residual or previously unresected tumor
* Willingness to undergo surgery and sign informed consent
* Patients not currently eligible for an alternate competing interventional clinical trial
* Enrollment in the Mayo Clinic Cancer Center Neuro-Oncology Program Registry for the study of Nervous System Tumors (IRB#12-003458)

Exclusion Criteria:

* Age < 18 years
* Found to be a member of a vulnerable population (e.g. pregnant, lacking capacity to consent) during the course of pre-enrollment or pre-surgical assessment
* Prior gross total resection of brain tumor leading to absence of visible latent disease (exemption available for post-operative enrollment)
* Any contraindication to surgery, including anyone who in the opinion of the surgeon is at unreasonably elevated risk of wound complications
* Patients who have not yet undergone surgery or radiation, but who would be appropriate candidates for an alternate interventional clinical trial (e.g. post-operative fractionated vs single fraction radiation to the surgical cavity for surgical brain metastases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of surgical resection by short and long term outcomes | Up to 5 years
  Feasibility will be evaluated by meeting enrollment criteria.
Incidence of adverse events | Up to 5 years
  Safety will be evaluated by recording adverse events utilizing proper reporting measures.

SECONDARY OUTCOMES:
Overall survival | Time from initial diagnosis to the date of death/or censored at the time of last known alive, assessed up to 5 years
  Median time of survival along with 95% confidence interval will be estimated using the Kaplan-Meier method.
Progression free survival | Time from initial diagnosis to the date progression is identified, assessed up to 5 years
  Median time of progress-free survival along with the 95% confidence interval will be estimated using the Kaplan Meier method.
Neurosurgical morbidity | Up to completion of surgery
  Postoperative complications such as wound infection and neurologic deficits will be logged. Additional metrics including hospital stay and readmission rates will also be logged. Standard descriptive statistics will be used to summarize the outcomes.
Time to subsequent treatment (i.e. chemotherapy/immunotherapy and/or radiation) | Time from surgical resection at Mayo Clinic until an adjuvant treatment is administered, assessed up to 5 years
  Median time to subsequent treatment along with the 95% confidence interval will be estimated using standard descriptive statistics.
Rate of local recurrence | Up to 5 years
  Will be logged as a categorical value and continuous data - endpoint is diagnosis of local recurrent disease. The presence and time to local recurrent disease will be logged and standard descriptive statistics will be used to summarize the outcomes.
Rate of leptomeningeal disease | Up to 5 years
  Will be logged as both a categorical value and continuous data - endpoint is diagnosis of leptomeningeal disease. The presence and time to occurrence of leptomeningeal disease will be logged and standard descriptive statistics will be used to summarize the outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Terry C. Burns, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials